CLINICAL TRIAL: NCT01753440
Title: Study on the Safety and Efficacy of Allogeneic Mesenchymal Stem Cell Implantation Combined With Bypass Grafting in Patients With Coronary Artery Disease and Ischemic Cardiomyopathy.
Brief Title: Allogeneic Stem Cells Implantation Combined With Coronary Bypass Grafting in Patients With Ischemic Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Kyriakos Anastasiadis, Professor Kyriakos Anastasiadis, AHEPA University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEPA_CTL_01
Record Dates: First submitted 2012-12-18; First posted 2012-12-20 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease; Ischemic Cardiomyopathy
Keywords: coronary artery disease; heart failure; stem cells implantation
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure | interventions — Inosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem cells implantation (Other): Patients with severe coronary artery disease and chronic ischemic cardiomyopathy with a LVEF ≤40% who are scheduled for elective CABG according to accepted guidelines. Additional criteria include the following: age <75 years, history of myocardial infarction (not less than 14 days before the procedure), LVEF ≤40 % assessed with echocardiography, and a distinct area of dyskinetic or akinetic left ventricular myocardium corresponding with the infarct localization.
  Interventions: Procedure: Intramyocardial implantation of of a novel mesenchymal precursor cell type (iMP).

INTERVENTIONS:
Procedure: Intramyocardial implantation of of a novel mesenchymal precursor cell type (iMP). — Intramyocardial implantation of a novel mesenchymal precursor cell type (iMP).

SUMMARY:
The aim of the present study is to investigate safety and efficacy of intramyocardial implantation of a novel mesenchymal precursor cell type (iMP) in patients with ischemic cardiomyopathy at the time of coronary artery bypass grafting.

DETAILED DESCRIPTION:
This study aims to investigates in situ cardiac regeneration utilizing precision delivery of a novel mesenchymal precursor cell type (iMP) during coronary artery bypass surgery (CABG) in patients with ischemic cardiomyopathy (LVEF < 40 %). Preoperative scintigraphy imaging (SPECT) will be used to identify hibernating myocardium not suitable for conventional myocardial revascularization for iMP implantation. iMP cells will be implanted intramyocardially in predefined viable peri-infarct areas that show poor perfusion, which could not be grafted due to poor target vessel quality. Postoperatively, SPECT will be used to identify changes in scar area.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years
* Severe coronary artery disease amenable to surgical revascularization according to current guidelines
* History of acute myocardial infarction at least 14 days previously
* Left ventricular ejection fraction (LVEF) ≤ 40% as assessed with echocardiography
* Distinct area of dyskinetic or akinetic left ventricular myocardium corresponding with the infarct localization
* Patient's informed consent obtained

Exclusion Criteria:

* Emergency operation
* Debilitating chronic disease (eg. malignancy or terminal renal failure)
* Concomitant valve surgery
* Previous cardiac surgery
* Malignant ventricular arrhythmias
* Haematologic disease
* Woman in reproductive age
* Severe psychiatric illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
iMP-related adverse events | 12 months
  Major adverse cardiac and cerebrovascular events including death, postoperative myocardial infarction, need for revascularization, stroke, hospitalization for worsening heart failure, myocardial rupture, infectious myocarditis, or sustained ventricular arrhythmias.
Hypersensitivity | 12 months
  Hypersensitivity reaction (fever, urticaria, hemolytic anemia, hypotension, immune thrombocytopenia)

SECONDARY OUTCOMES:
Scar reduction | 4 months
  Myocardial scar size reduction assessed with SPECT
Scar reduction | 12 months
  Myocardial scar size reduction assess with SPECT
LVEF | 12 months
  Left ventricular ejection fraction
Change in quality of life | 12 months
  Quality of life evaluated with MLHFQ

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, MD, PhD FETCS, Principal Investigator — AHEPA University Hospital
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Hare JM, Fishman JE, Gerstenblith G, DiFede Velazquez DL, Zambrano JP, Suncion VY, Tracy M, Ghersin E, Johnston PV, Brinker JA, Breton E, Davis-Sproul J, Schulman IH, Byrnes J, Mendizabal AM, Lowery MH, Rouy D, Altman P, Wong Po Foo C, Ruiz P, Amador A, Da Silva J, McNiece IK, Heldman AW, George R, Lardo A. Comparison of allogeneic vs autologous bone marrow-derived mesenchymal stem cells delivered by transendocardial injection in patients with ischemic cardiomyopathy: the POSEIDON randomized trial. JAMA. 2012 Dec 12;308(22):2369-79. doi: 10.1001/jama.2012.25321. PMID 23117550
- [Background] Anastasiadis K, Antonitsis P, Doumas A, Koliakos G, Argiriadou H, Vaitsopoulou C, Tossios P, Papakonstantinou C, Westaby S. Stem cells transplantation combined with long-term mechanical circulatory support enhances myocardial viability in end-stage ischemic cardiomyopathy. Int J Cardiol. 2012 Mar 22;155(3):e51-3. doi: 10.1016/j.ijcard.2011.07.062. Epub 2011 Aug 17. No abstract available. PMID 21852003
- [Background] Menasche P. Cardiac cell therapy: lessons from clinical trials. J Mol Cell Cardiol. 2011 Feb;50(2):258-65. doi: 10.1016/j.yjmcc.2010.06.010. Epub 2010 Jun 30. PMID 20600097